CLINICAL TRIAL: NCT06395896
Title: The Effect of Breast Cancer Prevention Journey Program on Women's Health Beliefs Towards Breast Cancer: Quasi Experimental Study
Brief Title: The Effect of Breast Cancer Prevention Journey Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nurbanu Odacı (Other Government)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Nurbanu Odacı, Lecturer, Lokman Hekim University
Organization: Lokman Hekim University (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LokmanHekimU-Hem-NO-01
Record Dates: First submitted 2024-04-28; First posted 2024-05-02 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer Female
Keywords: Breast Neoplasms; Health Belief Model; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: There are two groups: experimental group and control group.
Who Masked: Outcomes Assessor
Masking Description: The statistical evaluation will be performed by a person other than the researchers and the experimental and control groups will be anonymized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast Cancer Prevention Journey Program Group (Experimental): Participants will first receive structured "The Fighting Breast Cancer" training based on the Health Belief Model. Then they will be taken to mammography screening with a free transportation service and will be screened for cancer.
  Interventions: Other: Breast Cancer Prevention Journey Program Group
- Routine Cancer Screening Program Group (Other): Participants in the control group will not receive any additional intervention. This group will only receive routine intervention within the scope of the breast cancer screening program conducted by the Ministry of Health.
  Interventions: Other: Routine Cancer Screening Program Group

INTERVENTIONS:
Other: Breast Cancer Prevention Journey Program Group — The researcher will invite individuals to the study at Necip Fazıl Family Center and conduct a pre-test application. The day and time for the "Fight Against Breast Cancer" training, which is structured based on the Health Belief Model prepared by the researchers, will be determined and announced to the participants. The training will be held in a single session of 45-60 minutes. Slide presentation and a breast model showing the symptoms of breast cancer will be used as training materials. At the end of the training, it will be announced that free shuttle service will be provided for mammography screening and individuals will be invited to screening. On the specified day and time, participants will be taken to the "Cancer Early Diagnosis, Screening and Education Center (KETEM)" in Mamak and mammography screening will be performed. After the screening, a post-test will be performed.
  Arms: Breast Cancer Prevention Journey Program Group
Other: Routine Cancer Screening Program Group — Participants in the control group will not receive any additional intervention. This group will only receive routine intervention within the scope of the breast cancer screening program conducted by the Ministry of Health. Health Ministry of Türkiye offers free mammography screening for breast cancer to women over the age of 40. In this context, women are called to the centers by phone and mammography screening is performed free of charge.
  Arms: Routine Cancer Screening Program Group

SUMMARY:
The aim of this quasi-experimental study is to determine the effect of the "Breast Cancer Prevention Journey Program" on health beliefs about breast cancer in women over 40 years of age who have never had a mammogram before. The research aims to answer the following basic questions:

-Do women who participated in the "Breast Cancer Prevention Journey Program" have different health beliefs about breast cancer than women who did not participate in the program? The researchers will compare the program with routine care to see if the "Breast Cancer Prevention Journey Program" works. The study will be conducted in a quasi-experimental design with a pre-test post-test control group.

Participants in the experimental group will first participate in the "The fight against breast cancer" training structured according to the Health Belief Model. One week after the training, the participants in the experimental group will be taken to mammography screening with free shuttles.

Participants in the control group will not receive any additional intervention. This group will only receive routine intervention within the scope of the breast cancer screening program conducted by the Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 40-69
* Having never had a mammogram before

Exclusion Criteria:

* Being diagnosed with breast cancer
* Having had a breast operation

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Champion's Health Belief Model Scale in Breast Cancer Screening | two week
  This scale was developed to assess women's breast cancer beliefs (1984) and adapted into Turkish in 2004 (2004). It has a total of 52 items. It is a 5-point Likert-type scale. No single total score is obtained from the scale. The 8 sub-dimensions of the scale and the minimum and maximum scores that can be obtained are as follows; "Perception of sensitivity (min:3; max:15)", "Perception of severity (min:6; max:30)", "Perception of health motivation (min:5; max:25)", "Perception of benefit of breast self-examination (BSE) (min: 4; max:20)", 'Perception of benefit of breast self-examination (CBM) (min:10; max:50)', 'Barriers to CBM (min:8; max:40)', 'Perception of benefit of mammography (min:5; max:25)' and 'Barriers to mammography (min:11; max:55)'. Scale subscale scores are calculated by summing the scores. An increase in score is associated with a positive attitude in all sub-dimensions except the barrier sub-dimension. The Cronbach's Alpha value of the scale is between 0.69 and 0.83.

CONTACTS AND LOCATIONS:
Overall Officials: Nurbanu Odacı, Master, Principal Investigator — Lokman Hekim Universty
Locations (1):
- Lokman Hekim Üniversitesi, Ankara, Çankaya, Turkey (Türkiye)